CLINICAL TRIAL: NCT05614011
Title: Q-POC SARS-CoV-2 Assay (Q27001) Clinical Performance Study Plan
Brief Title: Q-POC SARS-CoV-2 Assay COVID-19 Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QuantuMDx Group Ltd (Industry)
Collaborators: New Day Diagnostics (Network); PathAI (Industry); Bright Research Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QVTP-39
Record Dates: First submitted 2022-11-10; First posted 2022-11-14 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical study enrolling adult patients with signs and symptoms that are consistent with SARS-CoV-2. Positive and negative specimens will be run on the Q-POC SARS-CoV-2 Assay in comparison with an FDA-approved reference standard to calculate both the positive percent agreement (PPA, or sensitivity) and the negative percent agreement (NPA, or specificity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Subjects 18+ years of age (Experimental): A healthcare professional will take a sample per subject for the comparator test, following the manufacturer's (IFU) in one nostril. Mid-turbinate swab samples will be taken from the opposite nostril using Copan FLOQ Swabs and placed into MSwab buffer (Q14-116-P02), for the candidate test. In instances where opposite nostrils cannot be swabbed for both the comparator and the test under investigation, a 15-minute wait period to allow for viral reloading must occur between collecting both the comparator and the test samples on the same nostril.
  Comparator RT-PCR samples will be shipped overnight with ice packs and processed for testing within 48 hours of collection. Candidate test samples will tested as soon as possible following collection, however if time is required between specimen collection and testing, the samples must be stored at 2-8 °C for up to 24 hours. Test samples must also be stored at 2-8 °C whilst the Q-POC test is running.
  Interventions: Diagnostic Test: RT-PCR Test; Diagnostic Test: Real-time PCR Test

INTERVENTIONS:
Diagnostic Test: RT-PCR Test — High sensitivity RT-PCR COVID-19 Test. A healthcare professional will take a sample per subject for the comparator test, following the manufacturer's Instructions For Use (IFU) in one nostril.
Diagnostic Test: Real-time PCR Test — Mid-turbinate nasal swab samples will be taken from the opposite nostril that was not swabbed for the comparator sample using Copan FLOQ swabs and placed into MSwab buffer. In instances where opposite nostrils cannot be swabbed for both the comparator and the candidate tests, a 15-minute waiting period to allow for viral reloading will occur before collecting the candidate test sample.
  Other Names: Q-POC

SUMMARY:
Q-POC SARS-CoV-2 moderate complexity PCR test performance evaluation

DETAILED DESCRIPTION:
The Q-POC SARS-CoV-2 Assay is a real-time PCR test intended for use on the Q-POC instrument for the qualitative detection of nucleic acids from Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), in nasal mid-turbinate swabs (MTSW) obtained from individuals suspected of COVID-19 by their healthcare provider. Testing is limited to laboratories certified under the Clinical Laboratory Improvement Amendments of 1988 (CLIA), 42 U.S.C. §263a, that meet requirements to perform high complexity or moderate complexity tests.

The Q-POC SARS-CoV-2 Assay is intended for use by laboratory personnel who have received specific training on the use of the Q-POC SARS-CoV-2 Assay in conjunction with the Q-POC instrument (Q29001).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 years.
* Participants must present with symptoms indicative of SARS-CoV-2 infection, within 0-5 days of symptom onset.
* Participants must have capacity to give informed consent.

Exclusion Criteria:

* Participant is under the age of 18 years.
* Participant does not have symptoms of SARS-CoV-2 infection.
* Participant lacks capacity to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Neilson, Study Director — QuantuMDx Group Ltd; Jason Liggett, PhD, Principal Investigator — New Day Diagnostics
Locations (3):
- United States (3):
  - Bright Research Center, Miami, Florida
  - EDP Biotech, Knoxville, Tennessee
  - PathAI, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects 18+ Years of Age: A healthcare professional will take a sample per subject for the comparator test, following the manufacturer's (IFU) in one nostril. Mid-turbinate swab samples will be taken from the opposite nostril using Copan FLOQ Swabs and placed into MSwab buffer (Q14-116-P02), for the candidate test. In instances where opposite nostrils cannot be swabbed for both the comparator and the test under investigation, a 15-minute wait period to allow for viral reloading must occur between collecting both the comparator and the test samples on the same nostril.
Period: Overall Study
Arm/Group | Subjects 18+ Years of Age
Started | 877
Completed | 877
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects 18+ Years of Age
Number analyzed (Participants) | 877
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 727
  >=65 years | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 560
  Male | 317
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0
  Asian | 7
  Black or African American | 358
  White | 62
  Hispanic/Latino | 43
  Other/Multiple Selections | 386
  Do Not Wish To Disclose | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 877

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Results on Both the Q-POC SARS-CoV-2 Assay and the RT-PCR Comparator Test
Description: The acceptance criteria for this study is Positive Percent Agreement (PPA) greater than or equal to 95% in a comparison between the Q-POC SARS-CoV-2 assay and the RT-PCR comparator test results
Time Frame: One hour
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects 18+ Years of Age
Number analyzed (Participants) | 877
Participants | 130

2. Primary Outcome: Number of Participants With Negative Results on Both the Q-POC SARS-CoV-2 Assay and the RT-PCR Comparator Test
Description: The acceptance criteria for this study is a Negative Percent Agreement (NPA) greater than or equal to 98% in a comparison between the Q-POC SARS-CoV-2 assay and the RT-PCR comparator test results.
Time Frame: One hour
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects 18+ Years of Age
Number analyzed (Participants) | 877
Participants | 736

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Subjects 18+ Years of Age
All-Cause Mortality (participants affected / at risk) | 0/877
Serious Adverse Events (participants affected / at risk) | 0/877
Other Adverse Events (participants affected / at risk) | 0/877

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT05614011/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT05614011/ICF_002.pdf